CLINICAL TRIAL: NCT05002959
Title: Retrospective and Prospective, Multicenter Study on T.E.S.S.® V3 (Implants and Instrumentation)
Brief Title: TESS V3 Modular Total Shoulder System PMCF
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2019-44E
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis Shoulder; Rheumatoid Arthritis; Rheumatoid Arthritis Shoulder; Avascular Necrosis; Revision; Rotator Cuff Tears; Osteonecrosis; Rotator Cuff Tear Arthropathy; Proximal Humeral Fracture; Malunion of Fracture, Shoulder Region
Keywords: Shoulder arthroplasty; Medical device; Performance; Safety; Shoulder prosthesis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteonecrosis; Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy; Shoulder Fractures; Fractures, Malunited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- TESS Anatomic: Subjects who received the Anatomic T.E.S.S.® V3 Modular Total Shoulder System to relieve pain and restore the joint function and who met the inclusion/exclusion criteria.
  Interventions: Device: Anatomic TESS V3
- TESS Reverse: Subjects who received the Reverse T.E.S.S.® V3 Modular Total Shoulder System to relieve pain and restore the joint function and who met the inclusion/exclusion criteria.
  Interventions: Device: Reverse TESS V3

INTERVENTIONS:
Device: Anatomic TESS V3 — Implantation of the T.E.S.S.® V3 Modular Total Shoulder System, Anatomic configuration.
  Groups: TESS Anatomic
Device: Reverse TESS V3 — Implantation of the T.E.S.S.® V3 Modular Total Shoulder System, Reverse configuration.
  Groups: TESS Reverse

SUMMARY:
This is a multicenter, retrospective and prospective, non-controlled post market surveillance study. The objectives of this study are to confirm safety, performance and clinical benefits of the T.E.S.S.® Version 3 Anatomic and Reverse Modular Total shoulder prosthesis and its instrumentation.

DETAILED DESCRIPTION:
The T.E.S.S.® (Total Evolutive Shoulder System) was developed to provide, with one instrumentation, a complete solution for all indications for shoulder arthroplasty: centered and eccentric rheumatoid osteoarthritis, necrosis, proximal fracture and mal-union of the humeral head. The T.E.S.S.® Modular system can be used in anatomic or reverse configurations with or without the use of a stem, providing a solution for hemi-arthroplasty, total shoulder arthroplasty and revision. The same instrumentation allows implantation of all versions of the T.E.S.S.®.

A maximum of 5 study centers will be involved in Europe. A total number of 146 implants, 73 T.E.S.S.® anatomic and 73 T.E.S.S.® reverse, will be included into the study. Each clinical site will be allowed to enroll a maximum 88 patients (60% of the total study cohort). Ethics Committee (EC) approval has to be obtained prior to conducting this study. All potential subjects will be required to participate in an informed consent process and sign the EC approved written informed consent prior to study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older and skeletally mature
* Patient is capable of understanding the surgeon's explanations and following his instructions, able and willing to participate in the follow-up program
* Patient gave consent to take part in the study by signing the Informed Consent Form
* Patient operated from January 2013 and received the Anatomic or Reverse T.E.S.S.® V3 Modular Total Shoulder System to relieve pain and restore the joint function
* Patient has adequate quality and quantity of bone stock to support the prosthesis
* Patient meets at least one of the following indications:

For anatomic type:

* Centered osteoarthritis of the shoulder
* Humeral head fractures
* Rheumatoid arthritis (with intact rotator cuff)
* Avascular necrosis of the humeral head
* Revision of a hemi-arthroplasty with a total arthroplasty
* Revision of a reverse prosthesis with an anatomic prosthesis
* Revision to increase the size of the stem (length and/or diameter)
* Revision of a glenoid prosthesis, a glenoid insert or a competitor's prosthesis

For reverse type:

* Offset osteoarthritis of the shoulder
* Massive and non-repairable rotator cuff tears
* Rheumatoid arthritis (with degenerative rotator cuff)
* Revision of an anatomic prosthesis with a reverse prosthesis
* Revision to increase the size of the stem (length and/or diameter)
* Revision of a glenoid prosthesis, a glenoid insert or a competitor's prosthesis

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program
* Patient is known to be pregnant or breastfeeding
* Patient has any condition that would, in the judgment of the Investigator, place the patient at undue risk or interfere with the study
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant)
* Patient who displays any of the following contra-indications cannot be included in this study:

  * Local or systemic infections
  * Severe muscular, neurological, or vascular deficiency of the affected joint
  * Poor bone quality likely to prevent osseointegration or to affect the long-term stability of the implant (Paget's disease, osteoporosis)
  * Any concomitant conditions likely to affect the function of the implant
  * Allergy to any of the implant components
  * Do not use the modular humeral version (screwed connection) in cases where the corolla cannot be two-thirds covered with bone stock and including the screwed modular stem/corolla junction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received a T.E.S.S.® Version 3 Anatomic or Reverse shoulder prosthesis from January 2013, based on the Indications for Use and who meet all of the inclusion and none of exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Implant survival at 10 years | 10 years
  The functional performance and clinical benefits will be determined by assessing the survival of the implant at 10 years using the Kaplan-Meier method. The survivorship of the implanted device will be recorded from the date of implantation to the date of revision or intended revision up to 10 years post-operatively.
Frequency and incidence of adverse events | 10 years
  The safety will be assessed by monitoring the frequency and incidence of adverse events.
  Adverse events will be collected in an Adverse Event Form, which gathers information on the date of occurrence, the nature of the adverse event, whether the device was involved, which treatment was used and the treatment outcome.

SECONDARY OUTCOMES:
Constant and Murley score | 10 years
  The functional performance and clinical benefits will be assessed by the Constant and Murley score.
  The Constant Murley score is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
EQ-5D-5L questionnaire | 10 years
  The functional performance and clinical benefits will be evaluated by collecting the patient-filled EQ-5D-5L questionnaire.
  EQ-5D-5L is a standardized instrument for measuring the health-related quality of life, which assesses health status in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each question has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to), which are singularly rated and then combined into a health status score, with higher scores indicating higher health utility. The second part of the EQ-5D-5L questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Radiographic Evaluation | 10 years
  The functional performance and clinical benefit will be evaluated by analyzing the post-operative radiographic parameters (radiolucency, osteolysis, osteophytes, component migration and heterotopic ossification). At each post-operative follow-up visit, the radiographies will be evaluated and any finding will be collected in a Radiographic Evaluation Form.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (2):
- France (2):
  - Lyon Ortho Clinic, Lyon
  - Clinique Saint-Jean (Group ORTHOSUD), Saint-Jean-de-Védas